CLINICAL TRIAL: NCT02860611
Title: Comparison of Th1 Cytokine Levels Between Type 1 and Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Gonca Incemehmet Tamer, Assoc. Professor, Istanbul Medeniyet University
Other Study IDs: IstanbulMU
Record Dates: First submitted 2016-08-04; First posted 2016-08-09 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes
Keywords: Type 1 diabetes; Type 2 diabetes; T helper 1 cytokines
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Type 1 Diabetes: Patients with type 1 diabetes
- Type 2 Diabetes: Patients with type 2 diabetes
- Control: Healthy volunteers

SUMMARY:
Recent reports show increased prevalence of obesity in patients with type 1 diabetes (T1DP)s while some studies stated that patients with type 2 diabetes (T2DPs) have islet cell auto-antibodies. These results raise the question of a common pathway in T1DM and T2DM via an association with T helper cells. In this study investigators aimed to investigate the difference between T helper 1 (Th1) cytokines levels in T1DPs, T2DPs and healthy subjects.

The study included 114 T1DPs on insulin treatment, 35 newly diagnosed T2DPs who had not used oral antidiabetics but insulin before and 31 healthy subjects (CG).

Serum interferon gamma (IFN-γ), interleukin-2 (IL-2) and tumor necrosis factor alpha (TNF-α) levels were measured using ELISA method. Serum levels of those cytokines in T1DPs were compared with those in T2DPs and controls.

ELIGIBILITY:
Inclusion Criteria:

* Being >18 years old
* Giving consent to participate

Exclusion Criteria:

* Acute and chronic inflammatory diseases
* significant concomitant disease likely to interfere with glucose metabolism,
* malignancies,
* hemoglobinopathies,
* In addition, glucose intolerance (fasting glucose level and that after glucose load) and HbA1C ≥ 5.7 % were also used exclusion criteria in the control group, group as American Diabetes Association (ADA) defined prediabetes as HbA1C between 5.7-6.4% (Standards of medical care in diabetes -2012. Diabetes care. 2012:35.)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study included 114 T1DPs on insulin treatment, 35 newly diagnosed T2DPs who had not used oral antidiabetics but insulin before and 31 healthy subjects (CG).
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2013-02; Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Difference in T helper cytokines between groups | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gonca Tamer, Principal Investigator — Istanbul Medeniyet University
Locations (1):
- Medeniyet University Goztepe Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No